CLINICAL TRIAL: NCT00684528
Title: A Double-Blind, Randomized, Active-Comparator (Metformin) Controlled, Clinical Trial to Study the Efficacy and Safety of the Strategy to Start Patients With Type 2 Diabetes Mellitus on Janumet™ Compared to Metformin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: jfr_il0801
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Type 2
Keywords: DM 2; Metformin; Januvia; Community setting; newly diagnosed diadetics, or diabetes patients not treated during the last year
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a (Active Comparator): This group will receive Metformin and placebo.
  Interventions: Drug: Metformin 1500 mg daily
- 2 (Experimental): The second arm will receive Metformin and Januvia
  Interventions: Drug: Metformin 1500 mg daily; Drug: Metformin + Janufer (Janumet)

INTERVENTIONS:
Drug: Metformin 1500 mg daily — 500 mg thrice daily
Drug: Metformin + Janufer (Janumet) — Titration up to 1500/150 mg daily
  Arms: 2

SUMMARY:
Comparison between the effectiveness of one anti-diabetic drug (Metformin, To combination of this drug and additional drug (Janufer), In the community setting.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-comparator (metformin) controlled study in drug-naïve patients with T2DM who have an HbA1c ≥ 7.5%. The duration of the study is 55 weeks, which will include a 1-week screening period (Visit 1 to Visit 2) and a 54 week double-blind, active treatment period. At Visit 2/Day 1 patients who meet all enrollment criteria will be randomized in a 1:1 ratio to one of two active treatment groups: 1. JANUMET™ (fixed-dose combination sitagliptin/metformin) or 2. metformin. The starting fixed-dose combination of sitagliptin/metformin will be 50/500 mg administered twice-daily and then up-titrated to a dose of 50/1000 mg b.i.d. over 4 weeks. The starting dose of metformin will be 500 mg twice-daily and then up-titrated to a dose of 1000 mg b.i.d. over 4 weeks. Patients who can not tolerate JANUMET™ at a dose of at least 50/500 mg b.i.d. or metformin at a dose of at least 500 mg b.i.d. 6 weeks after randomization and throughout the study will be discontinued. During the double-blind treatment period patients will remain on the study medication, but investigators are allowed to add other antihyperglycemic agents to improve glycemic control as necessary. The investigator can schedule additional visits to initiate additional antihyperglycemic agents or monitor glycemic control at any time during the study period. There will be no fixed visit schedule, but 7 clinical visits are recommended. It is also recommended to perform the first visit on active treatment 6 weeks after randomization and after this visit to schedule visits every 3 months. All clinical and lab data can be obtained using the "Clalit health care information system".

ELIGIBILITY:
Inclusion Criteria:

* All laboratory measurements are to be performed after an overnight fast ≥ 10 hours in duration. Patients with laboratory screening values/findings not meeting protocol inclusion criteria may, at the discretion of the investigator, have one repeat determination performed. If the repeat value satisfies the criterion they may continue in the screening process. Only the laboratory test not meeting inclusion should be repeated (not the entire panel).

Exclusion Criteria:

Glucose Metabolism and Therapy Criteria

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis. Patients Requiring Specific Treatments
* Patient has symptomatic hyperglycemia requiring immediate initiation of insulin therapy.
* Patient has a history of intolerance or hypersensitivity to metformin or sitagliptin or has any contraindication to use metformin.

Concomitant Disease of Organs and Systems

* Patient has a medical history of active liver disease (excluding hepatic steatosis).
* Patient has severe active peripheral vascular disease (e.g., manifested by claudication with minimal activity, a non-healing ischemic ulcer, or disease which is likely to require intervention such as with bypass or angioplasty).
* Patient has unstable or acute congestive heart failure.
* Patient has a history of malignancy without documentation of remission/cure. Other Criteria
* Patient is pregnant, has a positive urine pregnancy test at Visit 1, is expecting to conceive within the projected duration of the study, or is breast feeding.

Exclusion Criteria Based on Lab Abnormalities

* Patient has increased serum-creatinine and/or decreased estimated creatinine clearance.
* If screening labs are repeated, the last laboratory draw/result should be used for inclusion.§ Either elevated Creatinine or decreased estimated creatinine clearance lead to exclusion of the patient.
* Patients whose serum creatinine does not meet the exclusion criteria, but whose estimated creatinine clearance is <60 mL/min but ≥50 mL/min, may have a measured creatinine clearance (i.e., based upon a 24-hour urine collection). These patients may be eligible if their measured creatinine clearance is ≥60 mL/min.

At Visit 2

* Patient has a site fingerstick glucose <130 mg/dL (7.2 mmol/L) or >320 mg/dL (17.8 mmol/L).

Note: If the patient meets this exclusion criterion AND the investigator believes that the value does not reflect the patient's recent glycemic control based upon recent SBGM values and/or the Visit 1 FPG value, the patient should not be excluded at this time. The current visit should be changed to an "Unscheduled visit" and the patient should be rescheduled for Visit 2. If, at the rescheduled Visit 2, the patient meets this exclusion criterion, the patient MUST be excluded.

* Patient has a positive urine pregnancy test.
* Patient developed a new medical condition, suffered a change in status of an established medical condition, developed a laboratory abnormality, or required a new treatment or medication between Visit 1 and Visit 2 which meets any previously described study exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy and safety of community based study in diabetic patients, comparing Metformin to Metformin + Janufer. | 54 weeks
The efficacy and safety of Metformin VS Metformin + Janufer in the community setting | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Joel Zinger, MD, Principal Investigator — clali health organization
Locations (1):
- Clalit Health services center, Tel Aviv, Israel

REFERENCES:
- [Background] Mistry GC, Maes AL, Lasseter KC, Davies MJ, Gottesdiener KM, Wagner JA, Herman GA. Effect of sitagliptin, a dipeptidyl peptidase-4 inhibitor, on blood pressure in nondiabetic patients with mild to moderate hypertension. J Clin Pharmacol. 2008 May;48(5):592-8. doi: 10.1177/0091270008316885. Epub 2008 Mar 19. PMID 18353996
- [Result] Scott R, Loeys T, Davies MJ, Engel SS; Sitagliptin Study 801 Group. Efficacy and safety of sitagliptin when added to ongoing metformin therapy in patients with type 2 diabetes. Diabetes Obes Metab. 2008 Sep;10(10):959-69. doi: 10.1111/j.1463-1326.2007.00839.x. Epub 2008 Jan 14. PMID 18201203